CLINICAL TRIAL: NCT00080184
Title: Effectiveness of EEG Biofeedback in the Treatment of Fibromyalgia
Brief Title: Effectiveness of Brainwave Biofeedback in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000930-01A2 (NIH)
Record Dates: First submitted 2004-03-24; First posted 2004-03-25 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Electroencephalograph (EEG) biofeedback; Electromagnetic stimulation; Neurofeedback; Neurotherapy; Complementary and Alternative Medicine
MeSH Terms: conditions — Fibromyalgia

INTERVENTIONS:
Procedure: Low Energy Neurofeedback System

SUMMARY:
The purpose of this study is to determine whether a new form of brainwave biofeedback is effective in the treatment of fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a chronic disorder that involves chronic widespread musculoskeletal pain typically accompanied by fatigue, disordered sleep, cognitive complaints, psychological distress, and impairments in functioning. Treatments to date have been only partially effective and typically of modest benefit. Many persons with FM remain persistently dysfunctional and often disabled. This has given greater impetus for patients to seek complementary and alternative medicine (CAM) therapies. In this study, a variant of electroencephalograph (EEG) biofeedback known as Low Energy Neurofeedback System (LENS) will be used to reduce FM symptoms.

Participants in this study will be randomly assigned to receive either LENS or placebo for several sessions. The Fibromyalgia Impact Questionnaire will be used to assess participants at the end of the study and at the 3- and 6- month follow-up visits.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of fibromyalgia with symptoms for at least 1 year
* Self-report of having attention/concentration, memory, multi-tasking or other thinking difficulties
* Able to read and understand English
* Able to attend treatment sessions weekly and return for planned follow-ups
* Appropriate balance of average delta (<4 Hertz) EEG waveband and alpha (approximately 4-8 Hertz) EEG waveband amplitude on LENS screening (to be determined by study personnel);

Exclusion criteria:

* Other chronic pain condition of major significance
* Current chronic viral infection
* Current other unstable medical condition
* History of spinal, including neck, surgery
* Psychological screening indicates psychotic, suicidal, homicidal, and/or substance abusing
* Use of long-acting opioid medication taken on a continuous 24-hour dosing schedule
* Current involved in litigation regarding pain condition or seeking disability
* History of electroconvulsive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-12; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Mueller HH, Donaldson CC, Nelson DV, Layman M. Treatment of fibromyalgia incorporating EEG-Driven stimulation: a clinical outcomes study. J Clin Psychol. 2001 Jul;57(7):933-52. doi: 10.1002/jclp.1060. PMID 11406805